CLINICAL TRIAL: NCT06985901
Title: Evaluation of the Efficacy of Pulmonary Vein Isolation by Pulsed-field Ablation in Persistent Atrial Fibrillation: a Multicenter Study With Follow-up by Implantable Cardiac Monitor
Acronym: PersAF ICM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-API-03
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-06

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptomatic persistent atrial fibrillation (Experimental)
  Interventions: Procedure: Persistent atrial fibrillation ablation using Pulsed-field ablation

INTERVENTIONS:
Procedure: Persistent atrial fibrillation ablation using Pulsed-field ablation — Pulmonary vein isolation with pulsed-field ablation coupled with 3D electroanatomic mapping. Follow-up with insertable cardiac monitor.

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia in adult population. According to current guidelines for the management of AF, radiofrequency (RF) ablation (including at least pulmonary vein isolation [PVI]) is a validated therapeutic option for persistent AF. Recently, Pulsed-field ablation (PFA) - a new non-thermal energy - has been used to treat paroxysmal and persistent AF with a high success rate in observational studies. This new technology is based on tissue-specificity on myocardium, avoiding collateral damages on adjacent structures. Before confirming a superiority of PFA over existing thermal energies, prospective studies concerning an exclusive population of persistent AF patients are needed, with rigorous assessment of the recurrences using continuous monitoring (insertable cardiac monitor [ICM]). PFA efficacy using ICM has never been evaluated. Before considering PFA in therapeutic strategies through large-scale randomized studies using rigorous monitoring of recurrences, preliminary studies are needed in a persistent AF population-only. This pilot cohort study will provide solid data of PFA efficacy (using continuous monitoring of recurrences) for future randomized studies.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent AF (continuous episode sustained beyond 7 days)
* Refractory, intolerant or unwilling to take ADT
* Signed informed consent
* Affiliation to medical social coverage.

Non inclusion Criteria:

* Persistent long-term atrial fibrillation with ongoing episode continuous for more than 3 years;
* Left ventricular ejection fraction ≤ 15% ;
* Stage IV of the New York Heart Association classification;
* Previous atrial ablation outside the cavotricuspid isthmus;
* Wearer of an implantable electronic cardiac prosthesis (pacemaker or defibrillator; MCI)
* Hypertrophic heart disease other than hypertensive hypertrophic heart disease;
* Severe valvular heart disease, including the presence of a mechanical mitral valve or any mitral surgery;
* Congenital heart disease, including atrial septal defect, patent foramen ovale treated by percutaneous closure with atrial septal prosthesis;
* Presence of cardiac thrombus;
* Myocardial infarction or percutaneous coronary angioplasty within the last 6 months;
* Cardiac surgery within the last 6 months;
* Systemic thromboembolic event less than 6 months ago;
* Pulmonary embolism less than 6 months ago or pulmonary hypertension requiring specific treatment;
* Inability to read independently
* Vulnerable patient: minor, patient under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To assess the 12 month-efficacy (absence of atrial arrhythmias recurrences based upon ICM follow-up) after PVI using PFA in patients with persistent AF. | 12 months
  Efficacy will be assessed by the absence of AF/AT (episodes > 2min) recurrences during a 12-month follow-up period (clinical success) based upon continuous monitoring (ICM). Recurrence will be defined as any AF/AT episode > 2 min (detected by ICM) after the 2-month blanking period.

SECONDARY OUTCOMES:
Quantify the total atrial arrhythmias burden (AF/AT) over a 12-months period | 12 months
  Efficacy will be assessed by total AF/AT burden (recurrence as defined in the main criterion of evaluation), recorded by the ICM, and defined as the total period of time spent in AF/AT over the 12-month follow-up period (after the 2-month blanking period; assessment period of 10 months)
Assess patient distribution according to residual arrhythmias burden after one year | 12 months
  Residual AF/AT burden will be categorized into 4 groups: 0-0,1%; >0,1%-1%; >1-10%; >10% of the follow-up period. After calculation of the total AF/AT burden of each patient at M12, he will be classified into one of the above categories.